CLINICAL TRIAL: NCT01923506
Title: Stereotactic Body Radiation Therapy to the Prostate Fossa: Phase I Dose Escalation Study
Brief Title: Stereotactic Body Radiation Therapy in Treating Patients With Prostate Cancer After Undergoing Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13257; NCI-2013-01613 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 13257 (Other: City of Hope Medical Center)
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (SBRT) (Experimental): Patients receive 5 fractions of SBRT over 1.5 weeks.
  Interventions: Radiation: stereotactic body radiation therapy; Procedure: quality-of-life assessment; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — Undergo SBRT
  Other Names: SBRT; stereotactic radiation therapy; stereotactic radiotherapy
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of stereotactic body radiation therapy in treating patients with prostate cancer after undergoing surgery. Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) with an upper limit of 45 Gray (Gy) in 5 fractions, in the delivery of stereotactic body radiation therapy (SBRT) to the prostate fossa.

SECONDARY OBJECTIVES:

I. To assess acute and late toxicities from treatment.

II. To assess biochemical progression-free survival.

III. To collect prospective quality-of-life data related to bowel, urinary, and sexual health.

OUTLINE: This is a dose-escalation study.

Patients receive 5 fractions of SBRT over 1.5 weeks.

After completion of study treatment, patients are followed up at 90 days and then periodically for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* History of diagnosis of prostate cancer after undergoing prostatectomy
* No evidence of regional nodal or distant metastases based on computed tomography (CT) abdomen and pelvis and whole body bone scan within 120 days prior to study entry; nodes less than 1.5 cm will be considered reactive and biopsy is not required; nodes 1.5 cm or larger are required to undergo biopsy and be negative prior to study registration; bone scan findings in the absence of blastic or lytic lesion correlates on CT imaging will also be deemed non-neoplastic
* Eastern Cooperative Oncology Group (ECOG) performance scale 0-2
* Child bearing potential: In this patient population, this pertains to the ability to conceive a child; eligible patients already have received prostatectomy, and therefore this risk is not applicable
* Prostate specific antigen (PSA) value can be undetectable up to a value of 2.0 within 30 days prior to study entry
* PSA value that is undetectable can be enrolled if pathology from prostatectomy demonstrates one or more of the following: positive margin, extracapsular extension, or seminal vesicle invasion
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Patients should not have any uncontrolled illness including ongoing or active infection
* Patients may not be receiving any other investigational agents, or concurrent biological chemotherapy
* Patients with history of prior malignancies (with exception to non-melanoma skin cancer) are ineligible for this study, unless they are documented to be disease-free for at least 5 years
* Study-specific exclusions:

  * History of prior radiation to the pelvis
  * History of uncontrolled inflammatory bowel disease
  * Unable to comply with radiation therapy procedures
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-11-25 (Actual); Primary Completion 2026-07-28 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
MTD, defined as the highest dose tested in which fewer than 33% of patients experienced dose limiting toxicity, graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 90 days
  Tables will be created to summarize these toxicities and side effects by dose level.

SECONDARY OUTCOMES:
Incidence of acute toxicities observed at each dose level graded according to the NCI CTCAE version 4.0 | Up to 90 days
  Tables will be created to summarize these toxicities and side effects by dose level.
Incidence of late toxicities observed at each dose level graded according to the NCI CTCAE version 4.0 | Up to 3 years
  Tables will be created to summarize these toxicities and side effects by dose level.
Biochemical progression-free survival | Up to 3 years
  Estimated using Kaplan-Meier. 95% confidence intervals should be provided.
Prospective quality-of-life data related to bowel, urinary, and sexual health using the numerical scores generated from the patient questionnaires | Up to 3 years
  Quality of life questionnaires include the International Prostate Symptom Scale (IPSS), sexual health inventory for men (SHIM), and Merrick rectal function scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sagus Sampath, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States